CLINICAL TRIAL: NCT00604591
Title: Investigation of the Dopamine System in Frontotemporal Dementia
Brief Title: Effects of Tolcapone on Frontotemporal Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAF4151; 5R00NS060766 (NIH)
Record Dates: First submitted 2008-01-19; First posted 2008-01-30 (Estimated); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Frontotemporal Lobar Degeneration
Keywords: Dementia Treatment; Frontotemporal Dementia; Dopamine; Frontotemporal Lobar Degeneration
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Frontotemporal Dementia | interventions — Tolcapone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo then Tolcapone (Placebo Comparator): Participants take placebo during study week 1 and then tolcapone during week 3.
  On Day 1, 100 mg of tolcapone/placebo will be taken at three specific times: once in the morning, once in the afternoon, once at night. Then, from Days 2-6, 200 mg of tolcapone/placebo will be taken three times a day: once in the morning, once in the afternoon, once at night. On Day 7, 200 mg of tolcapone/placebo will be taken only in the morning and afternoon. On Day 8, 200 mg of tolcapone/placebo will be taken only in the morning. After the last dose on Day 8 is taken, the wash-out period begins and lasts through Day 14.
  Interventions: Drug: Tolcapone; Drug: Placebo
- Tolcapone then Placebo (Experimental): Participants take tolcapone during study week 1 and then placebo during week 3.
  On Day 1, 100 mg of tolcapone/placebo will be taken at three specific times: once in the morning, once in the afternoon, once at night. Then, from Days 2-6, 200 mg of tolcapone/placebo will be taken three times a day: once in the morning, once in the afternoon, once at night. On Day 7, 200 mg of tolcapone/placebo will be taken only in the morning and afternoon. On Day 8, 200 mg of tolcapone/placebo will be taken only in the morning. After the last dose on Day 8 is taken, the wash-out period begins and lasts through Day 14.
  Interventions: Drug: Tolcapone; Drug: Placebo

INTERVENTIONS:
Drug: Tolcapone — 200 mg by mouth three times a day
  Other Names: Tasmar
Drug: Placebo — 200 mg by mouth three times a day
  Other Names: Sugar pill

SUMMARY:
This study will test the effects of a medication called tolcapone on cognitive, behavioral, and language problems seen in patients with frontotemporal dementia (FTD). Tolcapone increases the amount of dopamine, a brain chemical that may be lowered in FTD. The study will see if tolcapone can improve thinking, behavior, and language in people with FTD and will look at the effects of the drug on brain activity.

Patients with FTD who are between 40 and 85 years of age may be eligible for this study.

Participants will be seen as outpatients at the Columbia University Medical Center approximately one a week for 4 weeks. They take tolcapone or a placebo (a look-alike pill with no active ingredient) during study week 1. During study week 3, those who took placebo during week 1 now take tolcapone for 1 week and those who took tolcapone now take placebo. In addition, patients undergo the following tests and procedures:

* Neurological tests to evaluate attention, problem-solving and memory. These tests are repeated several times during the course of the study.
* Test to look for a gene that affects the amount of dopamine in the brain, using blood samples collected in a previous study.
* Blood draws four times during the study.
* Functional MRI (fMRI) to learn about changes in brain regions that are involved in performing tasks. For fMRI, the patient lies on a table that can slide in and out of the scanner, a narrow metal cylinder surrounded by a magnetic field. The procedure takes about 60 minutes and is performed four times over the course of the . FMRI involves taking pictures of the brain during MRI while the subject performs a task so that changes in the brain that occur during these tasks can be studied.

DETAILED DESCRIPTION:
FTD is a significant cause of disability and death with an estimated prevalence of 15 cases per 100,000 persons in the 45- to 64-year-old age range. Despite the magnitude of this problem, there is currently a relative lack of understanding of the causes of, and treatments for, FTD, possibly because criteria for its diagnosis have only recently been developed. As an outcome of the proposed investigations, the investigators expect to determine the effects of cortical dopamine augmentation in FTD, evaluate the effect of dopamine augmentation on processing efficiency with fMRI, and explore the effects of a genetic polymorphism on symptom presentation and disease course. The research proposed in this protocol is significant because it could provide a new class of treatments for FTD, identify the fMRI findings associated with symptom improvement, and determine the contribution of a genetic polymorphism to symptom presentation and disease course.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of frontotemporal dementia (FTD)
* Age 40 to 85
* Assigned durable power of attorney
* Caregiver willing and able to accept the responsibilities involved in the study
* Mattis Dementia Rating Scale-2 (MDRS2) score less than 132

Exclusion Criteria:

* The diagnosis of any other type of dementia besides FTD including Alzheimer's disease, Lewy body dementia, vascular dementia, dementia associated with Parkinson's disease, corticobasal syndrome, and progressive supranuclear palsy.
* Known allergy or serious adverse reaction to tolcapone
* Active liver disease
* Current alcohol abuse
* Active substance abuse
* Elevated liver function tests
* Patient is taking tolcapone or any other catechol-O-methyltransferase (COMT) inhibitor, benserazide, alpha-methyldopa, dobutamine, apomorphine, isoproterenol, an monoamine oxidase inhibitor (MAO-I), or clozapine
* Symptomatic cardiovascular disease (e.g., angina, transient ischemic attack (TIA) , syncope)
* Uncontrolled hyper- or hypotension
* Any other contraindication to tolcapone
* Any medication that significantly affects the dopamine system, including stimulants and antipsychotic medications
* Pregnant women

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01-30 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2016-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Huey, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler CH, Singer C, O'Brien C, Hauser RA, Lew MF, Marek KL, Dorflinger E, Pedder S, Deptula D, Yoo K. Randomized, placebo-controlled study of tolcapone in patients with fluctuating Parkinson disease treated with levodopa-carbidopa. Tolcapone Fluctuator Study Group III. Arch Neurol. 1998 Aug;55(8):1089-95. doi: 10.1001/archneur.55.8.1089. PMID 9708959
- [Background] Apud JA, Mattay V, Chen J, Kolachana BS, Callicott JH, Rasetti R, Alce G, Iudicello JE, Akbar N, Egan MF, Goldberg TE, Weinberger DR. Tolcapone improves cognition and cortical information processing in normal human subjects. Neuropsychopharmacology. 2007 May;32(5):1011-20. doi: 10.1038/sj.npp.1301227. Epub 2006 Oct 25. PMID 17063156
- [Background] Baker M, Mackenzie IR, Pickering-Brown SM, Gass J, Rademakers R, Lindholm C, Snowden J, Adamson J, Sadovnick AD, Rollinson S, Cannon A, Dwosh E, Neary D, Melquist S, Richardson A, Dickson D, Berger Z, Eriksen J, Robinson T, Zehr C, Dickey CA, Crook R, McGowan E, Mann D, Boeve B, Feldman H, Hutton M. Mutations in progranulin cause tau-negative frontotemporal dementia linked to chromosome 17. Nature. 2006 Aug 24;442(7105):916-9. doi: 10.1038/nature05016. Epub 2006 Jul 16. PMID 16862116

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Tolcapone: Participants take placebo during study week 1 and then tolcapone during week 3. On Day 1, 100 mg of placebo will be taken at three specific times: once in the morning, once in the afternoon, once at night. Then, from Days 2-6, 200 mg of placebo will be taken three times a day: once in the morning, once in the afternoon, once at night. On Day 7, 200 mg of placebo will be taken only in the morning and afternoon. On Day 8, 200 mg of placebo will be taken only in the morning. After the last dose on Day 8 is taken, the wash-out period begins and lasts through Day 14.
- Tolcapone Then Placebo: Participants take tolcapone during study week 1 and then placebo during week 3.
  On Day 1, 100 mg of tolcapone will be taken at three specific times: once in the morning, once in the afternoon, once at night. Then, from Days 2-6, 200 mg of tolcapone will be taken three times a day: once in the morning, once in the afternoon, once at night. On Day 7, 200 mg of tolcapone will be taken only in the morning and afternoon. On Day 8, 200 mg of tolcapone will be taken only in the morning. After the last dose on Day 8 is taken, the wash-out period begins and lasts through Day 14.
Period: First Intervention (Day 1 to Day 8)
Arm/Group | Placebo Then Tolcapone | Tolcapone Then Placebo
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout (Day 9 to Day 14)
Arm/Group | Placebo Then Tolcapone | Tolcapone Then Placebo
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Second Intervention (Day 15 to Day 24)
Arm/Group | Placebo Then Tolcapone | Tolcapone Then Placebo
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Includes all participants who participated in the study since all participants received both tolcapone and placebo in this cross-over designed study. Participants were randomly assigned to start on tolcapone or placebo and then crossed over to received the alternative treatment after a wash-out period.
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Reaction Time on the N-back Cognitive Test [Mean (Standard Deviation); unit: milliseconds]
  0-back accuracy | 9141 (2225)
  1-back accuracy | 7863 (2323)

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time on the N-back Cognitive Test (0-back Condition)
Description: In the N-back task, subjects are given a response pad with response buttons numbered 1, 2, 3, and 4 at the points of a diamond-shaped box and shown a random series of numbers from 1 to 4 appearing for 500 ms every 1.8 seconds at locations corresponding to the positions of the numbers on the response pad. Instructions presented on the screen above the diamond instruct patients to recall the stimulus seen "N" numbers previously. In the 0-back condition, the subjects are instructed to press the button with the number on the screen. Three blocks of 40 images will be administered during the working memory task for a total of 120 images.
Time Frame: First intervention: Day 8 and Second intervention: Day 21
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Placebo: Participants take 100 mg of the placebo orally three times a day during the first day and then 200 mg orally for the next six days. On the seventh day, participants take 200 mg placebo twice a day. On the eighth day, particpants take 200 mg placebo once.
- Tolcapone: Participants take 100 mg of the tolcapone orally three times a day during the first day and then 200 mg orally for the next six days. On the seventh day, participants take 200 mg tolcapone twice a day. On the eighth day, particpants take 200 mg tolcapone once.
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 28 | 28
milliseconds | 7935 (2563) | 8322 (1940)

2. Primary Outcome: Reaction Time on the N-back Cognitive Test (1-back Condition)
Description: In the N-back task, subjects are given a response pad with response buttons numbered 1, 2, 3, and 4 at the points of a diamond-shaped box and shown a random series of numbers from 1 to 4 appearing for 500 ms every 1.8 seconds at locations corresponding to the positions of the numbers on the response pad. Instructions presented on the screen above the diamond instruct patients to recall the stimulus seen "N" numbers previously. In the 1-back condition, the subjects are instructed to report the number presented one number back from the number displayed on the screen. Three blocks of 40 images will be administered during the working memory task for a total of 120 images.
Time Frame: First intervention: Day 8 and Second intervention: Day 21
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 28 | 28
milliseconds | 7060 (2475) | 8226 (2842)

3. Secondary Outcome: Score on Neuropsychiatric Inventory Questionnaire (NPI-Q)
Description: The NPI-Q is a retrospective caregiver/informant-based interview that assesses 12 neuropsychiatric symptom domains including delusions, hallucinations, agitation/aggression, depression, anxiety, euphoria/elation, apathy/indifference, disinhibition, irritability/lability, aberrant motor behaviors, night-time behavioral disturbances and appetite/eating disturbances. Each symptom within a domain are rated by the caregiver in terms of severity (1=mild to 3=severe). Total scores are calculated by adding the composite scores to obtain a score ranging from 0 (no symptoms, better outcome) to 36.
Time Frame: First intervention: Day 8 and Second intervention: Day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 28 | 28
score on a scale | 8.68 (4.83) | 8.21 (4.50)

4. Secondary Outcome: Score on the Repeated Battery for the Assessment of Neurological Status (RBANS) for Dementia
Description: The RBANS is a brief, individually administered test that captures multiple cognitive domains, including attention, language, visuospatial/constructional abilities, immediate memory, and delayed memory. Index scores range from 0 to 20 (better outcome) for each of the 5 domains tested and the composite scores are added to generated a total index score, which ranges from 0 to 100 (better outcome).
Time Frame: First intervention: Day 8 and Second intervention: Day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 28 | 28
score on a scale | 67.89 (17.66) | 66.57 (18.32)

5. Secondary Outcome: Score on the Clinical Global Impressions (CGI) Scale
Description: The CGI is often used in treatment studies as a proxy for global functioning and is a subjective score assigned by the treating physician that incorporates elements of illness severity, patient distress, patient impairment, and functioning. The CGI is given a numerical ranking each visit after the first, with 6=major worsening, 5=mild worsening, 4=no change, 3=mild improvement, and 2=major improvement. Scores range from a 2 (better outcome) to a 6 (worse outcome).
Time Frame: First intervention: Day 8 and Second intervention: Day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Tolcapone
Number analyzed (Participants) | 28 | 28
score on a scale | 4.14 (0.76) | 3.75 (0.65)

ADVERSE EVENTS:
Time Frame: Up to 3 years to track any events during study participation.
Groups:
- All Participants: Adverse events data were not collected per Arm, therefore adverse events cannot be reported per Arm.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 6/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=28)
Elevated liver enzymes (Hepatobiliary disorders) | 6 (6)
Nausea (General disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Headache (General disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Upset Stomach (Gastrointestinal disorders) | 2 (2)
Hyperactive Bowel Syndrome (Gastrointestinal disorders) | 2 (2)
Moderate fall (Injury, poisoning and procedural complications) | 2 (2)

LIMITATIONS AND CAVEATS:
A modified and simplified version of the N-back task was used because patients with FTD were incapable of performing the original version. Another limitation was the relatively brief duration of treatment conditions and washout.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes